CLINICAL TRIAL: NCT02455895
Title: A Multicenter Randomized, Double-Masked Study Comparing the Efficacy of Novabay iLid Cleanser Versus Vehicle on Ocular Skin Flora
Brief Title: Efficacy of iLid Cleanser (Avenova) Versus Vehicle on Ocular Skin Flora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CM-01-14
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Sebaceous Gland Diseases; Blepharitis
Keywords: Blepharitis
MeSH Terms: conditions — Sebaceous Gland Diseases; Blepharitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iLid Cleanser (Avenova) (Active Comparator): iLid Cleanser - applied 2 times per day for 10 days
  Interventions: Device: iLid Cleanser
- iLid Cleanser Vehicle (Placebo Comparator): iLid Cleanser Vehicle - applied 2 times per day for 10 days
  Interventions: Device: iLid Cleanser

INTERVENTIONS:
Device: iLid Cleanser — Application of iLid Cleanser to reduce bacterial load on the lid and lash margins
  Other Names: Avenova

SUMMARY:
This study is designed to evaluate the effect of Novabay iLid Cleanser, as compared to its Vehicle, on the ocular skin flora.

In the pre-randomization phase, subjects will receive a single application of open-label NovaBay iLid Cleanser.

In the randomization phase of Stages 1 and 2, subjects will self-treat with masked Investigational Product twice daily for ten (10) days.

DETAILED DESCRIPTION:
This is an adaptive design, randomized, double-masked, vehicle-controlled, multicenter, parallel group study with two treatment arms: NovaBay iLid Cleanser ("Cleanser") and Cleanser Vehicle ("Vehicle").

The study will be conducted in two Stages, each preceded by a pre-randomization phase. Randomization of Cleanser:Vehicle will be 1:1 and 2:1 in Stages 1 and 2 respectively.

In the pre-randomization phase for Stages 1 and 2, subjects who meet all inclusion and no exclusion criteria will be evaluated by clinical examination at a single visit prior to having ocular skin specimens taken before and after treatment with open-label Cleanser.

In the randomization phase for both Stages 1 and 2, subjects who meet all inclusion and no exclusion criteria will be randomized and evaluated at three visits:

* Visit 1: Screening, Day 1
* Visit 2: Day 11 (+2) End of Treatment (EOT)
* Visit 3: Day 18 (±2) Post Treatment Evaluation/Exit Subjects will have ocular skin specimens taken at Visit 1, Day 1. The specimens will be collected before and 20 minutes after the first application of the study Investigational Product performed by study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, at least 6 years of age.
* Must be eligible for a recommendation to use eye lid cleansing/scrubs for:

  * Signs of acute or chronic blepharitis, such as eye lid debris (sleeves, collorates, flakes, crusting) requiring eye lid cleansing/scrubs, and/or
  * Signs consistent with mild, moderate, or severe meibomian gland disease (MGD) such as dilated and blocked glands with inspissated secretions sluggish or stagnant upon expression.
* Must be able to read, understand and sign an informed consent form that has been approved by an Institutional Review Board/Ethics Committee. If subject is less than 18 years of age, the informed consent must be signed and dated by subject's legally authorized representative (parent or guardian). Assent to participate should also be obtained from subjects under 18 years of age if required by local regulation.
* Must agree to comply with the visit schedule and other requirements of the study. The parent or guardian must agree to ensure compliance of subjects less than 18 years of age.
* Must agree to remove contact lenses, if applicable, for 15 minutes before and after application of the study Investigational Product.
* Must agree for the duration of the study to refrain from use of makeup/cosmetic products used around the eye(s) such as eye liner, mascara, and/or shadow, foundation or powder. Use of such products is allowed if the eyelid skin area is avoided.

Exclusion Criteria:

* Presence of signs and symptoms of bacterial or allergic conjunctivitis or allergic dermatitis at the Day 1 Visit.
* Suspected fungal, viral, Chlamydia or Acanthamoeba infection based on clinical diagnosis.
* Visual acuity not correctable to 1.0 LogMAR or better (equivalent to Snellen 20/200) in either eye using either a Snellen or ETDRS chart.
* Use of any topical ocular medications including tear substitutes during study participation.
* Use of any preserved or non-preserved glaucoma medications during the 14 days prior to Visit 1 and anticipated use during study participation.
* Presence of nasolacrimal duct obstruction.
* Presence of a punctal plug in either eye.
* Any systemic or ocular disease or disorder, complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study.
* Presence of active inflammation and/or active structural change in the cornea, iris or anterior chamber at the Day 1 visit.
* Use of any topical ocular or oral antimicrobial agent within the 3 days prior to Day 1 visit.
* Use of topical ocular corticosteroids or non-steroidal topical ocular anti-inflammatories (NSAIDs), within 3 days prior to study entry and during the trial.
* Use of RESTASIS® (Cyclosporine Ophthalmic Emulsion) 0.05%) in either eye during the trial.
* Any current immunosuppressive disorder (e.g., HIV positive), or use of immunosuppressive therapy (including chemotherapy).
* Participation in any other investigational clinical study within 30 days prior to study enrollment.
* Any subject who is on staff at the investigational site or is a family member of staff personnel.
* Additionally, the Investigator or Medical Monitor may declare any subject ineligible for a sound medical reason.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-01 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Microbiological efficacy | 20 minutes after application of test article
  Quantitative assessment of numbers of recoverable bacteria before versus after application of test article

SECONDARY OUTCOMES:
Ocular Signs | Assessed on Visit 1(Day 1), Visit 2 (Day 11) and Visit 3 (Day 18)
  lid erythema, lid swelling, lid crusting and debris on lashes, bulbar and palpebral conjunctival injection, and meibomian gland secretions (after expression)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Stroman, Ph.D., Study Director — NovaBay Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Ophthalmic Research Consultants of Arizona, Phoenix, Arizona
  - Turner Eye Institute, San Leandro, California
  - James D. Branch, MD, Winston-Salem, North Carolina